CLINICAL TRIAL: NCT06927375
Title: Clinical Study on the Combined Use of Tocilizumab and Flupentixol-Melitracen in the Treatment of Thyroid-Associated Ophthalmopathy: A Prospective Exploratory Study
Brief Title: A Study on the Combined Use of Tocilizumab and Flupentixol-Melitracen in the Treatment of Thyroid-Associated Ophthalmopathy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, lu ying li, Chief physician，head of Endocrinology department, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH9H-2024-T313-2
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Thyroid-Associated Ophthalmopathy
Keywords: Thyroid Eye Disease; Graves Orbitopathy; Thyroid Associated Ophthalmopathy; TAO; TED
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — tocilizumab; flupentixol, melitracen drug combination; Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tocilizumab combined with Flupentixol Melitracen (Experimental)
  Interventions: Drug: Tocilizumab(400mg) combined with Flupentixol Melitracen(0.5mg:10mg)
- Tocilizumab (Active Comparator)
  Interventions: Drug: Tocilizumab(400mg)

INTERVENTIONS:
Drug: Tocilizumab(400mg) combined with Flupentixol Melitracen(0.5mg:10mg) — Tocilizumab (Actemra) is administered via intravenous infusion at a dose of 400 mg at Weeks 0, 4, and 8. Flupentixol/Melitracen is given orally at a dose of 0.5 mg/10 mg twice daily for 8 consecutive weeks starting from Week 0.
  Other Names: study group
  Arms: Tocilizumab combined with Flupentixol Melitracen
Drug: Tocilizumab(400mg) — Tocilizumab (Actemra) is administered via intravenous infusion at a dose of 400 mg at Weeks 0, 4, and 8.
  Other Names: control group
  Arms: Tocilizumab

SUMMARY:
Thyroid-associated ophthalmopathy (TAO) is a serious, progressive, vision-threatening autoimmune disease that can be categorized into mild, moderate, and severe stages based on severity. The activity of TAO is commonly evaluated using the Clinical Activity Score (CAS). Tocilizumab serves as a second-line treatment option for patients with moderate to severe active TAO. Additionally, it is common for TAO patients to experience anxiety, which may exacerbate their condition and negatively impact prognosis. Therefore, we have designed this randomized controlled study to evaluate the impact of Flupentixol Melitracen (Lepan) on the treatment outcomes of participants receiving Tocilizumab (Actemra).

DETAILED DESCRIPTION:
Thyroid-associated ophthalmopathy (TAO) is a serious, progressive, vision-threatening autoimmune disease with an incidence rate of about 19-42 per 100,000. Currently, it ranks first among orbital diseases and is one of the primary causes of blindness. The extensive involvement of intraorbital tissues and the significant variability in the course of moderate to severe active TAO make its treatment outcomes uncertain, classifying it as refractory thyroid-associated ophthalmopathy. The pathogenesis of TAO has not been fully elucidated; however, activation of the thyrotropin receptor (TSHR) and insulin-like growth factor receptor-1 (IGF-1R) complex is considered a critical step in TAO, leading to abnormal immune proliferation responses within the orbit, causing hypertrophy of extraocular muscles and increased orbital fat tissue. These changes result in various clinical manifestations such as exophthalmos, diplopia, pain, and compressive optic neuropathy. Intravenous glucocorticoid therapy is recommended as the first-line treatment by guidelines, yet this treatment often leads to numerous side effects (including Cushing's facies, elevated blood pressure, glucose, and lipid levels, osteoporosis, urinary tract infections, peptic ulcers, etc.), and many patients with moderate to severe active TAO do not show significant improvement in ocular symptoms (such as impairment of eye movement, blurred vision, diplopia, etc.). Therefore, scholars at home and abroad have been committed to finding new effective treatments for refractory TAO. Biological agents represent emerging therapies for TAO, with domestic and international multicenter randomized controlled trials confirming that tocilizumab is effective in treating TAO and can be considered as a second-line treatment option for moderate to severe active TAO. Tocilizumab is a monoclonal antibody against the IL-6 receptor. Interleukin-6 (IL-6) can activate T cells and B cells and produce TSHR-stimulating immunoglobulins, and it can also directly act on preadipocytes in the orbit to promote adipose hyperplasia. Tocilizumab reduces memory B cell and immunoglobulin levels, thereby improving eye movements and clinical activity scores (CAS), and enhancing quality of life scores.

Most TAO patients exhibit proptosis, and severe cases may develop incomplete eyelid closure, resulting in exposure keratitis, corneal ulcers, and significant eye pain, photophobia, and lacrimation. Changes in appearance due to TAO and even potential blindness can cause patients to experience significant psychological stress, leading to feelings of inferiority, anxiety, depression, and other negative emotions. Additionally, patients with coexisting hyperthyroidism may exhibit irritability, insomnia, anger, and other emotional reactions. Studies have shown that serum and tear fluid IL-6 levels are elevated in TAO patients, which are hormone factors related to behavioral and emotional changes and can influence emotional regulation, including anxiety modulation, by acting on the brain. Moreover, neurogenic inflammation is considered part of the psychosomatic pathogenic mechanism of TAO. Under conditions of prolonged anxiety and psychological stress, TAO patients release norepinephrine from primary neurons, generating neurogenic inflammation, and enhance the pro-inflammatory effects of platelets and leukocytes. Anxiety and depression levels in TAO patients are higher than those in other chronic diseases, increasing the risk of unnatural deaths, including suicide, thus impacting public health. Several studies indicate that TAO significantly affects patients' quality of life, including reduced participation in daily activities and poorer emotional health, and adverse emotions like anxiety and depression might exacerbate the condition and affect prognosis.

Therefore, while treating the symptoms of thyroid-associated eye disease, attention should also be paid to the varying degrees of negative psychology experienced by these patients, necessitating enhanced psychological interventions for them. We hypothesize that in refractory TAO patients with anxiety, combined treatment with Flupentixol Melitracen might help alleviate anxiety and depressive moods, improve quality of life, facilitate treatment, and improve ocular prognosis. This clinical study aims to evaluate the efficacy of tocilizumab (Actemra) in combination with Flupentixol Melitracen (Lepan) in the treatment of refractory thyroid-associated ophthalmopathy.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 80 years (inclusive).
* Meets internationally recognized diagnostic criteria for TED with the more severely affected eye in moderate to severe active phase. Meeting any one of the following criteria qualifies as moderate to severe: an exophthalmos ≥2 mm compared with normal values for sex and race; presence of inconstant to constant diplopia; a lid retraction ≥2 mm. A Clinical Activity Score (CAS) of ≥3 or a score of 2 combined with MRI evidence indicating active disease is defined as active.
* Normal thyroid function within one month prior to enrollment: including those currently taking antithyroid drugs or not requiring medication, with FT3 and FT4 levels within normal range and TSH either normal or decreased.
* HAMA (Hamilton Anxiety Rating Scale) score of ≥14.
* Voluntary participation and provision of informed consent.

Exclusion Criteria:

* Severe cardiac, hepatic, or renal insufficiency (including myocardial ischemia or myocardial infarction, arrhythmias, and heart failure; ALT, AST ≥ 3 times the upper limit of normal; eGFR < 60 ml/min/1.73 m²).
* communicable disease.
* Pregnancy or planning to become pregnant.
* Currently breastfeeding.
* Received radioactive iodine treatment or hepatitis vaccination within three months prior to enrollment.
* Received systemic immunotherapy for TAO, including oral or intravenous glucocorticoids, other immunosuppressants, or orbital radiotherapy within one month prior to enrollment.
* Planning to undergo other treatments during the course of this study.
* Severe mental disorders that affect compliance.
* Presence of other clinically significant or unstable systemic diseases.
* Patients who are unlikely to complete the entire course of treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-11-12 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
comprehensive score | week12
  The comprehensive score has a maximum of 30 points. It is calculated as follows：the half score of TED-QoL (Thyroid Eye Disease Quality of Life questionnaire) (15 points), plus the higher value of CAS (Clinical Activity Score) between the two eyes (7 points). Additionally, one point is added for each symptom present in the participant: tearing, photophobia, dry eye, blurred vision. Also included are diplopia score (3 points) and restricted eye movement score (1 point). The study investigates changes in the comprehensive score before and after treatment in two groups.

SECONDARY OUTCOMES:
Go-qol | week 12
  The change from baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire visual function score and psychosocial function score, and the total score.
TED-QoL | week 12
  The change from baseline in the TED-QoL.
CAS Decrease by ≥2 Points | week 12
  The proportion of participants whose higher CAS value decreased by ≥2 points compared to baseline.
CAS Change Value | week 12
  The change in CAS value compared to baseline for participants.
Diplopia Improvement | week 12
  The proportion of participants whose diplopia score decreased by ≥1 point.
Proptosis Change | week 12
  The change in proptosis (eye protrusion) compared to baseline for participants
overall response | week 12
  The proportion of participants who experience reduction of proptosis ≥2 mm and reduction of CAS ≥2 points
The comprehensive score of TED-QoL and CAS | week12
  The comprehensive score has a maximum of 14 points. It is calculated as follows：the 7/30 score of TED-QoL (Thyroid Eye Disease Quality of Life questionnaire) (7 points), plus the higher value of CAS (Clinical Activity Score) between the two eyes (7 points).The study investigates changes in the comprehensive score before and after treatment in two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yingli Lu, Study Chair — Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China; Qin Li, Principal Investigator — Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No